CLINICAL TRIAL: NCT01339208
Title: TREAT (Telemedicine for Reach, Education, Access, and Treatment)
Acronym: TREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda Siminerio, Director Diabetes Institute, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO10100547
Record Dates: First submitted 2011-04-14; First posted 2011-04-20 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2011-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telemedicine Diabetes Intervention (Experimental)
  Interventions: Other: Telemedicine diabetes intervention

INTERVENTIONS:
Other: Telemedicine diabetes intervention — 3 month duration telemedicine consultation and diabetes education

SUMMARY:
The purpose of this study is to evaluate the feasibility and clinical efficacy of an innovative care model that combines Telemedicine consultations, educator therapeutic management and diabetes education to empower patients to be in greater control of their own diabetes care for improvements in diabetes outcomes.

DETAILED DESCRIPTION:
This study will assess whether a new care delivery model combining telemedicine videoconference diabetes consultations with diabetes self-management teaching is efficacious in reducing HbA1c in patients with type 2 diabetes in rural areas. The control group will consist of patients with type 2 diabetes receiving "usual care", i.e., who have not received a referral to the endocrinologist telemedicine team. Secondary outcomes include patient satisfaction, level of understanding of self-management skills, and hypoglycemia

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older with type 2 diabetes
* Referral by a primary care provider.
* HbA1c equal or greater than 7.0%.

Exclusion Criteria:

* Type 1 diabetes
* Gestational Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c % from baseline | 3 and 6 month

SECONDARY OUTCOMES:
Patient satisfaction | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Frederico Toledo, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Northwest, Seneca, Pennsylvania, United States

REFERENCES:
- [Derived] Toledo FG, Ruppert K, Huber KA, Siminerio LM. Efficacy of the Telemedicine for Reach, Education, Access, and Treatment (TREAT) model for diabetes care. Diabetes Care. 2014 Aug;37(8):e179-80. doi: 10.2337/dc13-1909. No abstract available. PMID 25061149